CLINICAL TRIAL: NCT05301348
Title: In Vivo Detection of Circulating Clots in Patients With Thromboembolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 239347
Record Dates: First submitted 2022-02-09; First posted 2022-03-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Procedure (Experimental): Subjects will receive PAFC procedure
  Interventions: Device: Photoacoustic Flow Cytometry

INTERVENTIONS:
Device: Photoacoustic Flow Cytometry — Detection of circulating blood clots

SUMMARY:
Subjects with thromboembolic disease or at high-risk for thromboembolic conditions diagnosed with ultrasound or other standard of care techniques will be recruited to estimate the feasibility of a device to detect in vivo CBCs.

DETAILED DESCRIPTION:
There are no current gold standards to detect circulating blood clots. The sensitivity of most current methods to detect CBCs is poor when low numbers are present in the host. A novel method of detecting circulating blood clots, PAFC, may improve detection of CBCs and, if so, ultimately may reduce complications related to previously undetected clots.

ELIGIBILITY:
Inclusion Criteria

* Men and women, 18 years old and older.
* Evidence of current venous or arterial thromboembolic disease diagnosed by standard of care clinical, radiographic, or laboratory testing or acute ischemic stroke.
* Informed consent provided by the subject.

Exclusion Criteria

* Pulmonary embolus with a need for mechanical ventilation or other ventilator support (may be on oxygen delivered by nasal cannula or mask at an FiO2 of ≤ 0.40)
* Acute coronary syndrome (including unstable angina)
* Significant cardiac arrhythmia (may have atrial fibrillation controlled with medication)
* Intracardiac thrombus
* Any embolus or thrombus requiring vascular surgery or interventional radiology to attempt acute embolectomy or thrombectomy
* Sickle cell disease with vaso-occlusive crisis
* Sepsis or life-threatening infection
* Traumatic injury requiring hospitalization (within 30 days prior to enrollment)
* Pregnancy or breastfeeding
* Severe mental illness
* Other conditions deemed by the investigators to put the subject at greater risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Circulating blood clots detected by PAFC with D-dimer levels in patients with known venous thromboembolic disease - Positive PA peaks | 30 days
  Measurement of in vivo CBC-associated positive PA peaks in a signal trace of patients who have been diagnosed with conventional methods.
Comparison of Circulating blood clots detected by PAFC with D-dimer levels in patients with known venous thromboembolic disease - Negative PA peaks | 30 days
  Measurement of in vivo CBC-associated negative PA peaks in a signal trace of patients who have been diagnosed with conventional methods.

SECONDARY OUTCOMES:
Relationship between PA peaks and circulating blood clots | 30 days
  PAFC will be compared with the fibrin degradation fragment D-dimer to indicate the presence of a blood clot undergoing dissolution.
Safety of the PAFC method - skin sensitivity | 30 days
  The safety of the PAFC device through estimation of the sensitivity of the individual's skin to laser radiation will be indicated by a possible warming feeling or tingling sensation.
Safety of the PAFC method - change in skin property | 30 days
  The safety of the PAFC device through estimation of the change to the skin's property after laser exposure measured by appearance of possible red spots in the irradiated local area

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeeva Onteddu, MD, Principal Investigator — University of Arkansas; Jonathan A Young, Study Director — University of Arkansas
Locations (1):
- Univerisity of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dressler DK. Death by clot: acute coronary syndromes, ischemic stroke, pulmonary embolism, and disseminated intravascular coagulation. AACN Adv Crit Care. 2009 Apr-Jun;20(2):166-76. doi: 10.1097/NCI.0b013e3181a0b5e8. PMID 19411875
- [Background] Nedosekin DA, Sarimollaoglu M, Galanzha EI, Sawant R, Torchilin VP, Verkhusha VV, Ma J, Frank MH, Biris AS, Zharov VP. Synergy of photoacoustic and fluorescence flow cytometry of circulating cells with negative and positive contrasts. J Biophotonics. 2013 May;6(5):425-34. doi: 10.1002/jbio.201200047. Epub 2012 Aug 20. PMID 22903924
- [Background] Juratli MA, Menyaev YA, Sarimollaoglu M, Melerzanov AV, Nedosekin DA, Culp WC, Suen JY, Galanzha EI, Zharov VP. Noninvasive label-free detection of circulating white and red blood clots in deep vessels with a focused photoacoustic probe. Biomed Opt Express. 2018 Oct 23;9(11):5667-5677. doi: 10.1364/BOE.9.005667. eCollection 2018 Nov 1. PMID 30460154
- [Background] Cushman M. Epidemiology and risk factors for venous thrombosis. Semin Hematol. 2007 Apr;44(2):62-9. doi: 10.1053/j.seminhematol.2007.02.004. PMID 17433897
- [Background] Heit JA. Venous thromboembolism: disease burden, outcomes and risk factors. J Thromb Haemost. 2005 Aug;3(8):1611-7. doi: 10.1111/j.1538-7836.2005.01415.x. PMID 16102026
- [Background] Anderson FA Jr, Wheeler HB, Goldberg RJ, Hosmer DW, Patwardhan NA, Jovanovic B, Forcier A, Dalen JE. A population-based perspective of the hospital incidence and case-fatality rates of deep vein thrombosis and pulmonary embolism. The Worcester DVT Study. Arch Intern Med. 1991 May;151(5):933-8. PMID 2025141
- [Background] Juratli MA, Menyaev YA, Sarimollaoglu M, Siegel ER, Nedosekin DA, Suen JY, Melerzanov AV, Juratli TA, Galanzha EI, Zharov VP. Real-Time Label-Free Embolus Detection Using In Vivo Photoacoustic Flow Cytometry. PLoS One. 2016 May 26;11(5):e0156269. doi: 10.1371/journal.pone.0156269. eCollection 2016. PMID 27227413
- [Background] Galanzha EI, Sarimollaoglu M, Nedosekin DA, Keyrouz SG, Mehta JL, Zharov VP. In vivo flow cytometry of circulating clots using negative photothermal and photoacoustic contrasts. Cytometry A. 2011 Oct;79(10):814-24. doi: 10.1002/cyto.a.21106. Epub 2011 Aug 16. PMID 21976458
- [Background] Galanzha EI, Zharov VP. Photoacoustic flow cytometry. Methods. 2012 Jul;57(3):280-96. doi: 10.1016/j.ymeth.2012.06.009. Epub 2012 Jun 26. PMID 22749928